CLINICAL TRIAL: NCT03928613
Title: Efficacy of the Cognitive Training Based on Location Information and Activity in People With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Institute of Information & Communications Technology Planning & Evaluation, Korea (Unknown)
Responsible Party: Principal Investigator, Ji Won Han, Associate Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-1903-526-301
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognitive training; Cognitive intervention; Cognitive rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mild Cognitive Impairment (Experimental): * Clinical dementia rating 0 or 0.5
  * Diagnosed by physicians as mild cognitive impairment according to the criteria of International Working Group on Mild Cognitive Impairment
  Interventions: Behavioral: tablet based Cognitive Training based on location information

INTERVENTIONS:
Behavioral: tablet based Cognitive Training based on location information — Participants perform Tablet based Cognitive training using interactive voice services and tags three times (minimum 30 minutes per time) a week for 6 weeks

SUMMARY:
The purpose of this study is to examine therapeutic efficacy of cognitive Training based on location information and activity in people with mild cognitive impairment

DETAILED DESCRIPTION:
* A single arm, open-label study.
* Cognitive Training based on location information and activity is consists of both cognitive training and exercise(walking) using objects in the participant's home. The researchers visit the participant's home and find objects that were mainly used in the real life and easy to access (table, computer, television, etc.) and attach the recognition Bluetooth Low Energy(BLE) Tag (sticker integrated). The stickers printed on the tags consist of word categories (eg animals) belonging to a particular category, so as to assist strategic recall in the stepped recall task. The participants follow the instruction from the tablet-based program to perform the task. During performing the cognitive training program, the participants are guided to walk between the tagged objects in their home.
* The participants are aged over 60 years old and diagnosed with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 60
* Confirmed literacy o Diagnosed with mild cognitive impairment by International Working Group on Mild Cognitive Impairment and Clinical Dementia Rating(CDR) of 0 or 0.5.

Exclusion Criteria:

* Evidence of delirium, confusion
* Any neurological conditions causing cognitive decline such as Parkinson's disease, brain hemorrhage, brain tumor, normal pressure hydrocephalus
* Evidence of severe cerebrovascular pathology
* Presence of depressive symptoms that could influence cognitive function
* Presence of medical comorbidities that could result in any difficulties in study participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change in CERAD-TS1 score | baseline and 6 weeks
  Total Score of the Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Neuropsychological Assessment Battery (CERAD-TS1) . CERAD-TS1 is generated by simply summing the scores of six tests including the 1) Verbal fluency (range 0-24), 2) Boston naming test (0-15), 3) Word List Memory (0-30), 4) Word List Recall (0-10), 5) Word list recognition (0-10), 6) Constructional Praxis (0-11). The range of CERAD-TS1 score is 0 to 100 points), and the higher score represents the better cognitive function.

SECONDARY OUTCOMES:
Change in MMSE score | baseline and 6 weeks
  Mini-Mental State Examination (MMSE), ranged 0-30, the higher score represents the better cognitive function
Change in SMCQ score | baseline and 6 weeks
  Subjective Memory Complaint Questionnaire (SMCQ), ranged 0-14, the higher score represents the more difficulties in memory function for everyday life
Change in GDS score | baseline and 6 weeks
  Geriatric depression scale (GDS), ranged 0-30, the higher score represents the more severe depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ji Won Han, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital,, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No